CLINICAL TRIAL: NCT01739751
Title: Effect of a Program of Physical Activity Enhancement Using Pedometers in Chronic Obstructive Pulmonary Disease
Brief Title: Physical Activity Enhancement Using Pedometers in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Dr. Laura Mendoza, MD, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SA10i20022
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: COPD
Keywords: COPD; Physical activity; Pedometers; steps; non pharmacological treatment; rehabilitation; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients without feedback of a pedometers, followed for 3 months
- Pedometers (Experimental): With a program of physical activity enhancement using pedometers as a feedback
  Interventions: Device: pedometers

INTERVENTIONS:
Device: pedometers — portable device that estimate the number of steps walked daily
  Other Names: PD 724
  Arms: Pedometers

SUMMARY:
Physical activity is reduced in COPD affecting morbidity and mortality and the usual advice is not good enough to increase the physical activity level. The aim of the study is to determine the effects of pedometers in the physical level in COPD patients.

DETAILED DESCRIPTION:
Physical activity is reduced in COPD patients and has a negative effect in the morbidity and mortality of this condition. Unfortunately, usual advice is not good enough to reverse the sedentary condition in COPD patients. Pedometers are broadly used to measure and to enhance physical activity in COPD but their effects in COPD are not well known. The aim of the study is to determine the effects of a program using pedometers as a feedback in stable ex smokers COPD patients. Patients are recruited for a 3 months individual program promoting daily physical activity enhancement and are randomly assigned either to a pedometer-based program (experimental group) or to usual care (control group, the measurements at the beginning and at the end of the study are: anthropometrics, Spirometry, dyspnea, quality of life, exercise capacity and the average one week daily steps. Also the number of acute exacerbations during the follow up are recorded.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis according to GOLD guidelines
* Pack year Index equal or more than 10
* smoking suspended > 2 months
* older than 40 years old,

Exclusion Criteria:

* any chronic condition that does not allow walking
* participation in a rehabilitation program
* Acute exacerbation in the last two months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
effect in average steps walked daily | 3 months
  Comparison between both groups in the difference of the average of steps walked daily at final evaluation with the basal evaluation

SECONDARY OUTCOMES:
six minute walking distance | 3 months
  Comparison between groups in the difference of the distance( meters) in the six minute walking test in the final evaluation with the basal evaluation
score in the Saint George Respiratory Questionnaire | 3 months
  Comparison between groups in the difference of the score of the SGRQ at the final evaluation in comparison with the basal evaluation
Score of the COPD Assessment Test (CAT) | 3 months
  Comparison between groups in the difference of the CAT score at the final evaluation with the basal evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mendoza, MD, Principal Investigator — Hospital Clínico University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Bravata DM, Smith-Spangler C, Sundaram V, Gienger AL, Lin N, Lewis R, Stave CD, Olkin I, Sirard JR. Using pedometers to increase physical activity and improve health: a systematic review. JAMA. 2007 Nov 21;298(19):2296-304. doi: 10.1001/jama.298.19.2296. PMID 18029834